CLINICAL TRIAL: NCT03602573
Title: Nonalcoholic Fatty Liver Disease and Associated Liver Fibrosis in Peri-menopausal Women
Brief Title: Liver Fibrosis in Peri-menopausal Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Cheng Chen, Associate professor, Chang Gung Memorial Hospital
Other Study IDs: LSM-PMW
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Nonalcoholic Steatohepatitis; Liver Fibroses; Menopause
Keywords: Nonalcoholic steatohepatitis; Liver fibrosis; Menopause; Hormone
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre-menopause
- post-menopause

SUMMARY:
This is a prospective observational study in a single medical center.

The aim is to evaluate the status of fibrosis and steatosis of liver parenchyma in peri-menopausal women using noninvasive methods of vibration-controlled transient elastography (VCTE) with controlled attenuation parameter (CAP) and serum biomarkers.

Recruitment period: 2018/08/01 to 2019/07/31

Patient number: 200 females

Inclusion criteria:

1. Females, age of 46-55 years
2. Willing and able to comply with the study requirements
3. Willing and able to provide written informed consent to participate in the study

Exclusion criteria:

1. Unable to complete the noninvasive procedure of VCET and CAP
2. Unwilling to provide written informed consent to participate in the study

Laboratory tests and examinations:

Baseline and two follow-up visits (every 6 months):

1. Blood pressure
2. BW, BH, waist circumference, BMI
3. Complete blood cell (CBC) count
4. Albumin, AST, ALT, alkaline phosphatase, total bilirubin, r-GT, uric acid, hsCRP
5. Sugar (fasting), HbA1c, insulin, HOMA-IR
6. DM lipid profiles, adiponectin, leptin
7. Liver ultrasound, FibroScan touch 520
8. FSH, Estrodiol (E2), LH
9. TSH, free T4
10. HBsAg, anti-HCV, HBV DNA, HCV RNA, HBsAg quantification, HBV genotype (if HBsAg or anti-HCV positive)
11. ANA, Anti-mitochondrial antibody
12. Review history of drug and menstruation cycles

ELIGIBILITY:
Inclusion Criteria:

1. Females, age of 46-55 years
2. Willing and able to comply with the study requirements
3. Willing and able to provide written informed consent to participate in the study

Exclusion Criteria:

1. Unable to complete the noninvasive procedure of VCET and CAP
2. Unwilling to provide written informed consent to participate in the study

Ages: 46 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females, age of 46-55 years, premenopause and postmenopause
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
The impact of estrogen level on liver steatosis by FibroScan touch 520 | 1 year
  The association of estrogen level with the severity of liver steatosis.
The impact of estrogen level on liver fibrosis by FibroScan touch 520 | 1 year
  The association of estrogen level with the severity of liver fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Cheng Chen, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan